CLINICAL TRIAL: NCT03654898
Title: VITAL Start (Video-intervention to Inspire Treatment Adherence for Life): Brief Facility-based Video Intervention to Improve Retention and Adherence to ART Among Pregnant and Breastfeeding Women
Brief Title: VITAL Start: Brief Facility-based Video Intervention
Acronym: VITAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Maria Hyoun Kim, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H-39785; R01MH115793-01A1 (NIH)
Record Dates: First submitted 2018-08-23; First posted 2018-08-31 (Actual); Results first posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: HIV/AIDS
Keywords: pregnant women; viral suppression; retention; video intervention; pre-ART; counseling; HIV; adherence; PMTCT
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Investigators, Data analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VITAL Start (Active Comparator): VITAL Start: Video-based pre-ART counseling
  Interventions: Behavioral: VITAL Start: Video-based pre-ART counseling
- Standard of Care (Placebo Comparator): pre-ART education as conducted via routine facility methods
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: VITAL Start: Video-based pre-ART counseling — Patients in the experimental group will receive VITAL start pre-ARV counseling (approximately 27 minutes video followed by 10 minute guided Q & A to reinforce key messages and provide an opening for individual counseling=approximately total 37 minutes). This will be delivered by study staff.
  Arms: VITAL Start
Behavioral: Standard of Care — Patients randomized to the control arm will receive the usual standard of care (SOC) pre ARV initiation education with the National ARV Educational Flipchart
  Arms: Standard of Care

SUMMARY:
This a multi-center, parallel group, randomized controlled outcome assessor blinded trial with a qualitative descriptive component that seeks to assess the effectiveness of a brief facility-based video intervention to optimize retention and adherence to ART among pregnant and breastfeeding women with HIV infection.

DETAILED DESCRIPTION:
Universal HIV testing and treatment can accelerate population-level ART initiation and is critical to realize the UNAIDS 90-90-90 goals. Malawi pioneered Option B+ (B+), a novel application of test-and-treat that provided life-long ART for HIV+ pregnant and breastfeeding women. While maternal ART uptake improved 7-fold, retention and adherence remained suboptimal: only 59% were retained after two years, and of these, only two-thirds achieved adequate ART adherence. Other B+ countries are observing suboptimal retention.

VITAL Start (Video-intervention to Inspire Treatment Adherence for Life) is a brief facility-based video intervention, created with formative participatory research, applied theoretical frameworks, and evidence-based message framing techniques. VITAL Start was designed to help optimize retention and adherence to ART among pregnant and breastfeeding women in Malawi.

The study will evaluate the impact, implementation and cost effectiveness of VITAL Start in a multisite randomized controlled trial (RCT) in Malawi with the primary composite outcome of retention and adherence (viral suppression) 12 months after starting antiretroviral therapy (ART). The study will also examine the delivery of VITAL Start via surveys and interviews with patients and partners and conduct cost-effectiveness analyses.

If successful, VITAL Start will provide an intervention that (1) standardizes and improves counseling at a critical teaching moment through an engaging and culturally sensitive experience, (2) is inexpensive and rapidly scalable without decelerating ART expansion, and (3) allows more efficient use of health care worker time.

ELIGIBILITY:
Inclusion Criteria:

* Women who are HIV positive by two antibody rapid tests approved by the Malawi Ministry of Health
* Women age ≥18 years or 16-17 years if married or have a child
* Women who understand chichewa
* Women who are willing to provide informed consent
* Women who intend to remain in the health center catchment area for at least 6 months

Exclusion Criteria:

* Women already on ART
* Women with significant pre-existing psychiatric comorbidity at enrollment that may impact ability to provide consent according to the clinical judgment of study personnel (including cognitive impairment or known psychotic disorder)
* Women who participated in the study pilot

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Kim, MD, MSc, Principal Investigator — Baylor College of Medicine Childrens foundation Malawi
Locations (1):
- Baylor-Malawi, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: No
Data will be analysed by blinded study staff

REFERENCES:
- [Derived] Kim MH, Tembo TA, Mazenga A, Yu X, Myer L, Sabelli R, Flick R, Hartig M, Wetzel E, Simon K, Ahmed S, Nyirenda R, Kazembe PN, Mphande M, Mkandawire A, Chitani MJ, Markham C, Ciaranello A, Abrams EJ. The Video intervention to Inspire Treatment Adherence for Life (VITAL Start): protocol for a multisite randomized controlled trial of a brief video-based intervention to improve antiretroviral adherence and retention among HIV-infected pregnant women in Malawi. Trials. 2020 Feb 19;21(1):207. doi: 10.1186/s13063-020-4131-8. PMID 32075677

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | VITAL Start
Started | 395 (Two participants were disqualified after enrollment. Both were disqualified because they were already on ART. Therefore, the baseline characteristics for 393 participants are reported in this arm.) | 405 (Four participants were disqualified after enrollment. Reasons for disqualification were that women 1) were already on ART (n=2); 2) participated in the VITAL Start pilot (n=1); 3) not pregnant at follow-up ANC visit five weeks after study enrollment (n=1). Therefore, the baseline characteristics for 401 participants are reported in this arm.)
Completed | 304 | 314
Not Completed | 91 | 91

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | VITAL Start | Total
Number analyzed (Participants) | 393 | 401 | 794
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.08 (5.68) | 27.52 (5.67) | 27.30 (5.68)
Age, Customized [Count of Participants; unit: Participants]
  15-19 years | 28 | 21 | 49
  20-29 years | 245 | 247 | 492
  30-39 years | 114 | 125 | 239
  40 years or above | 6 | 8 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 393 | 401 | 794
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 393 | 401 | 794
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Education [Count of Participants; unit: Participants]
  No education | 17 | 22 | 39
  Some primary school (standard 1-5) | 108 | 83 | 191
  Primary completed (standard 6-8) | 114 | 135 | 249
  Some secondary (forms 1-2) | 72 | 78 | 150
  Secondary completed (forms 3-4) | 66 | 69 | 135
  Post-secondary | 16 | 14 | 30
Head of household [Count of Participants; unit: Participants]
  No | 320 | 330 | 650
  Yes | 73 | 71 | 144
Number of pregnancies [Count of Participants; unit: Participants]
  First | 55 | 62 | 117
  Second/third/fourth | 290 | 285 | 575
  More than four | 48 | 54 | 102
ART Regimen [Count of Participants; unit: Participants]
  DTG-based ART | 192 | 196 | 388
  EFV and other ART | 201 | 205 | 406

OUTCOME MEASURES:

1. Primary Outcome: Composite of Retention in ART Clinic and Viral Suppression
Description: This outcome is an aggregate measure. The study will measure if participants are both retained in ART clinic and also virally suppressed. Participants will be considered retained in care if they are verified by clinic records as active on ART. Amongst those retained the study will then assess viral suppression which will be measured as viral load less than 1,000 copies per milliliter.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | VITAL Start
Number analyzed (Participants) | 393 | 401
Participants | 206 | 220
Statistical Analysis 1: Comparison: Standard of Care vs VITAL Start; Test type: Superiority; p = 0.49, Chi-squared; cross-tabulation = 0.48
Statistical Analysis 2: Comparison: Standard of Care vs VITAL Start; Test type: Superiority; p = 0.67, Regression, Logistic; Adjusted logistic regression; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.80 to 1.42]

2. Secondary Outcome: Number of Participants With Good Self-reported Behavioral Adherence
Description: Self-reported adherence will be measured by a three-item adherence scale. The three items will include an assessment of the number of days with missed ART doses in the preceding 30 days; a scale rating of how good a job the participant did taking their medicines in the preceding 30 days and a scale rating of how often the participant took their medicines the way they were supposed to in the preceding 30 days. Item responses for the three adherence items will be linearly transformed to a 0-100 scale.
  Scores will be analyzed as a binary variable, with a score >/=90 good adherence and <90 not good adherence.
Time Frame: 12 months
Population: The outcome was assessed only among those who had a study visit at month 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | VITAL Start
Number analyzed (Participants) | 302 | 312
Participants | 248 | 248
Statistical Analysis 1: Comparison: Standard of Care vs VITAL Start; Test type: Superiority; p = 0.40, Chi-squared; Cross-tabulation = 0.71

3. Secondary Outcome: Number of Participants With Good (Daily) ART Adherence Was Measured by Drug Concentration in the Blood
Description: The concentration of two metabolites, Tenofovir diphosphate (TFVdp) and lamivudine triphosphate (3TCtp), was used to objectively measure ART adherence. The concentration of each metabolite was classified as low, medium, or high. TFVdp (low: <560; medium: 560 to 1399; and high: 1400 to 20900 fmol/sample) and 3TCtp (low: <400; medium: 400 to 799; and high: 800 to 2100 fmol/sample). For either metabolite, the high category suggests the participant had good (daily) ART adherence.
Time Frame: Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | VITAL Start
Number analyzed (Participants) | 293 | 299
Participants
  TFVdp: Low | 67 | 64
  TFVdp: Medium | 38 | 35
  TFVdp: High | 188 | 200
  3TCtp: Low | 130 | 115
  3TCtp: Medium | 122 | 138
  3TCtp: High | 41 | 46
Statistical Analysis 1: Comparison: Standard of Care vs VITAL Start; Test 1 was for TFVdp while test 2 was for 3TCtp; Test type: Superiority; p = 0.78, Chi-squared; Cross-tabulation = 0.50
Statistical Analysis 2: Comparison: Standard of Care vs VITAL Start; Test 2 was for 3TCtp while test 1 was for TFVdp; Test type: Superiority; p = 0.34, Chi-squared; Cross-tabulation = 2.13

ADVERSE EVENTS:
Time Frame: through study completion, an average of 1 year
Arm/Group | VITAL Start | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/405 | 3/395
Serious Adverse Events (participants affected / at risk) | 0/405 | 3/395
Other Adverse Events (participants affected / at risk) | 22/405 | 14/395
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VITAL Start (N=405) | Standard of Care (N=395)
Death (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Death (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VITAL Start (N=405) | Standard of Care (N=395)
Intimate partner violence and social harm (Social circumstances) | 22 | 14

LIMITATIONS AND CAVEATS:
1. Recruitment was slow due to the declining number of women living with HIV not already on ART at antenatal care clinics.
2. Recruitment was interrupted by the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT03654898/Prot_SAP_ICF_000.pdf